CLINICAL TRIAL: NCT02356276
Title: A Phase III Study of Hyperthermic Intraperitoneal Chemotherapy in the Treatment of Locally Advanced Gastric Cancer After radIcal Gastrectomy With D2
Brief Title: Efficacy of HIPEC in the Treatment of Locally Advanced Gastric Cancer After radIcal Gastrectomy With D2
Acronym: EHTLAGCRGD2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Zhejiang Cancer Hospital (Other); The Second Hospital of Hebei Medical University (Other); Chinese PLA General Hospital (Other); Henan Cancer Hospital (Other Government); Harbin Medical University (Other); Central South University (Other); Guangdong Provincial People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sun Yat-sen University (Other); Hebei Medical University Fourth Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-01
Record Dates: First submitted 2015-01-29; First posted 2015-02-05 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Gastric Cancer
Keywords: locally advanced gastric cancer; Hyperthermic Intraperitoneal Chemotherapy; radical gastrectomy with D2 lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIPEC group (Experimental): Postoperative hyperthermic intraperitoneal chemotherapy (HIPEC) is performed after radical surgery, followed by 6-8 cycles of systemic chemotherapy. The first HIPEC is conducted within 48 h after surgery: Paclitaxel 75 mg/m^2, 43°C, 60min. The second HIPEC is performed after 24 hours of the first HIPEC. The regimens are Paclitaxel 100 mg/m^2, 43°C, 60min.
  Systemic chemotherapy (XELOX or SOX regimens):
  XELOX regimen: Oxaliplatin: 130 mg/m^2, IV, d1; Capecitabine: 1 g/m^2 bid, days 1-14, every 3 weeks for a total of 6-8 cycles.
  If XELOX regimen is not conducted in some collaborators, SOX regimen is also permitted. The regimen is Oxaliplatin: 130 mg/m^2, IV, d1; S-1, 40-60 mg/m^2 bid, po, day 1-14, every 3 weeks for a total of 6-8 cycles.
  Interventions: Procedure: D2 lymphadenectomy; Procedure: Hyperthermic Intraperitoneal Chemotherapy; Drug: Systemic chemotherapy (XELOX or SOX regimens)
- Control group (Placebo Comparator): 6-8 cycles of systemic chemotherapy (XELOX or SOX regimens) were performed after radical gastrectomy with D2 lymphadenectomy.
  XELOX regimen is Oxaliplatin: 130 mg/m^2, IV, d1; Capecitabine: 1 g/m^2 bid, days 1-14, every 3 weeks for a total of 6-8 cycles.
  If XELOX regimen is not conducted in some collaborators, SOX regimen as comment systemic chemotherapy in Asia is also permitted to treat the patients. The treatment bundles are listed as follows: Oxaliplatin: 130 mg/m^2, IV, d1; S-1, 40-60 mg/m^2 bid (S-1: BSA <1.25m^2, 40mg bid, 1.25m^2≤ BSA ≤1.5m^2, 50mg bid, BSA>1.5m^2, 60 mg bid), po, day 1-14, every 3 weeks for a total of 6-8 cycles.
  Interventions: Procedure: D2 lymphadenectomy; Drug: Systemic chemotherapy (XELOX or SOX regimens)

INTERVENTIONS:
Procedure: D2 lymphadenectomy
  Other Names: surgical resection or radical surgery
Procedure: Hyperthermic Intraperitoneal Chemotherapy — The first HIPEC is conducted within 48 h after surgery: Normal saline 3000 -4000ml, Paclitaxel 75mg/m^2, 43°C, 60min. The second HIPEC is performed after 24 hours of the first HIPEC. The regimens are Paclitaxel 100 mg/m^2, 43°C, 60min.
  Other Names: HIPEC
  Arms: HIPEC group
Drug: Systemic chemotherapy (XELOX or SOX regimens) — XELOX regimen: Oxaliplatin: 130 mg/m^2, IV, d1; Capecitabine: 1 g/m^2 bid, days 1-14, every 3 weeks for a total of 6-8 cycles.
  SOX regimen: Oxaliplatin: 130 mg/m^2, IV, d1; S-1, 40 mg/m^2 bid, po, day 1-14 (S-1: BSA <1.25m^2, 40mg bid, 1.25m^2≤ BSA ≤1.5m^2, 50mg bid, BSA>1.5m^2, 60 mg bid) bid, d1-14, po, every 3 weeks for a total of 6-8 cycles.
  Other Names: XELOX or SOX regimens

SUMMARY:
HIPEC-01 is a prospective, open, randomized multicenter phase III clinical study conducted in China. To determine the efficacy of hyperthermic intraperitoneal chemotherapy (HIPEC) in the treatment of locally advanced gastric cancer, patients are randomized into HIPEC group and control group. In HIPEC group, the patients undergo radical gastrectomy with D2 lymphadenectomy and HIPEC with paclitaxel and postoperative chemotherapy. Patients in the control group just undergo radical gastrectomy with D2 lymphadenectomy followed by postoperative chemotherapy. Patients in both groups receive 6-8 cycles of postoperative systemic chemotherapy (XELOX or SOX regimens) and are followed up for 5 years or until death.

DETAILED DESCRIPTION:
Gastric cancer (GC) is the fourth most common cancer, and the second leading cause of cancer-related death worldwide. Advances in diagnostic and therapeutic approaches have achieved long-term survival for early GC. However, receiving perioperative/postoperative systemic chemotherapy and gastrectomy with D1-D2 lymph node dissection, 5-year survival rates of advanced gastric cancer remain under 30%. 40-60% of recurrences are peritoneal and/or locoregional. hyperthermic intraperitoneal chemotherapy (HIPEC) technique is increasingly used in the curative treatment of primary and digestive peritoneal carcinomatosis, in association with cytoreductive surgery. Theoretically, HIPEC eliminates free cancer cells that can be released into peritoneal cavity during the gastrectomy and prevents peritoneal carcinomatosis recurrences. The benefit of using HIPEC as an adjuvant treatment for advanced gastric cancer has been reported in several randomized studies and a meta-analysis. Surgical resection combined with HIPEC significantly reduces the peritoneal recurrences and improves the overall survival of GC patients. But there is not a prospective and randomized phase III clinical study of HIPEC in the treatment of locally advanced gastric cancer after radical surgery in China so far.

In order to evaluate the survival benefit and safety of radical surgery and HIPEC followed by postoperative chemotherapy in local advanced gastric cancer, patients who fulfill the inclusion and exclusion criteria will be recruited in this study and randomized to two treatment groups (HIPEC group and control group). In HIPEC group, the patients undergo radical gastrectomy with D2 lymphadenectomy and HIPEC with paclitaxel and postoperative chemotherapy. Patients in the control group just undergo radical gastrectomy with D2 lymphadenectomy followed by postoperative chemotherapy. Patients in both groups receive 6-8 cycles of postoperative systemic chemotherapy (XELOX or SOX regimens) . Patients are followed up for 5 years and the survival outcome will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 < age ≤ 70 years old
* Male or Non pregnant female
* The Eastern Cooperative Oncology Group (ECOG) status 0-1
* T3 or T4 gastric adenocarcinoma (visual determination according to AJCC 2010 7th edition)
* No distance metastasis, eligible for D2 lymphadenectomy
* Have not received cytotoxic chemotherapy, radiotherapy or immunotherapy
* White blood cells > 4,000/mm3
* neutrophils ≥ 1,500/mm3
* platelets ≥ 100,000/mm3
* hemoglobin>9g/l
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) < or = 2.5 times upper limit of nominal (ULN)
* total bilirubin (TBIL) < 1.5 times ULN
* serum creatinine < 1 times ULN
* Having given written informed consent prior to any procedure related to the study

Exclusion Criteria:

* Have other cancer within 5 years
* Existence of distance metastasis during surgey (M1)
* Prior malignant tumors with detectable signs of recurrence or distant metastasis
* Poorly controlled disease e.g. atrial fibrillation, stenocardia, cardiac insufficiency, persistent hypertension despite medicinal treatment, ejection fraction<50%
* Epileptic seizures patients need medicine control
* Uncontroled mental disease or mental disorder
* Drug abuse or psychological or social factors affect the judgment of results
* Contraindication to any therapy contained in this regimen specific to the study
* Receiving other chemotherapy, radiotherapy or immunotherapy
* Without given written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2015-05-11 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years
  assess overall survival during 5 years in both study arms

SECONDARY OUTCOMES:
5-year progression-free survival | 5 years
  assess progression-free survival rate during 5 years in both study arms
liver metastatic rate | 5 years
  calculate the percent of liver metastatic in both two arms during 5 years
local recurrence rate | 5 years
  calculate the percent of local recurrence in both two arms during 5 years
side effects | 5 years
  determine percent of adverse events or side effects according to NCI criteria, Common Terminology Criteria for AE (CTCAE 4.0).

OTHER OUTCOMES:
CEA mRNA expression of peritoneal lavage fluid | Through study completion, an average of 3 year
  Quantitative RT-PCR is used to analyze CEA mRNA expression of peritoneal lavage fluid before and after D2 lymphadenectomy between two arms

CONTACTS AND LOCATIONS:
Overall Officials: shuzhong cui, M.D, Study Director — Affiliated Tumor Hospital of Guangzhou Medical University Recruiting
Locations (14):
- China (14):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, China, Wuhan, Hubei
  - The second Xiangya Hospital of Central South University, Changsha, Hunan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hanzhou, Zhejiang